CLINICAL TRIAL: NCT02847273
Title: Peripheral Four-wavelength Near-infrared Spectroscopy Measurement: a Comparison Between EQUANOX and O3 in Cardiac Surgery
Acronym: NIRS-8
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0502
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Conventional Cardiac Surgery With Bypass
Keywords: NIRS; Regional oxygen saturation; cardiac surgery with bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Near-infrared spectroscopy (NIRS) is a continuous and non-invasive technology that measures regional tissue oxygen saturation (rSO2). Whatever the anatomical site of measurement, a normal value of rSO2 would suggest a good adequacy between oxygen supply and consumption at the regional level. Beside the trend ability of previous 2 or 3-wavelength devices, a new 4-wavelength generation of NIRS monitors which could reliably assess real-time absolute values of rSO2 is now available. The investigators aimed to compare peripheral absolute rSO2 values given by the 4-wavelength EQUANOX device 7600 (Nonin Medical, Plymouth, Mn) and the new O3 device (Masimo, Irvine, CA) during conventional cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Scheduled for conventional elective cardiac surgery with cardiopulmonary bypass
* Hospitalized in the Teaching University Hospital Louis Pradel (Lyon, France)
* Patient agreement

Exclusion Criteria:

* Age<18 years
* Black skin
* Emergencies
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Were included 20 caucasian adult patients scheduled for conventional elective cardiac surgery with cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Peripheral absolute rSO2 values | at conventional cardiac surgery (Day 1)
  Peripheral absolute rSO2 values given by the 4-wavelength EQUANOX device 7600 (Nonin Medical, Plymouth, Mn) and the new O3 device (Masimo, Irvine, CA) during conventional cardiac surgery.

SECONDARY OUTCOMES:
Arterial pressure | at conventional cardiac surgery (Day 1)
  General monitoring
heart rate | at conventional cardiac surgery (Day 1)
  General monitoring
pulse oxygen saturation | at conventional cardiac surgery (Day 1)
  General monitoring
bispectral index | at conventional cardiac surgery (Day 1)
  General monitoring
Inotrope drugs doses | at conventional cardiac surgery (Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Fellahi, Pr, MD PhD, Principal Investigator — Hôpital Cardiovasculaire et Pneumologique Louis Pradel, Hospices Civils de Lyon
Locations (1):
- Hôpital Cardiovasculaire et Pneumologique Louis Pradel, Hospices Civils de Lyon, Bron, France